CLINICAL TRIAL: NCT02477618
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of SAGE-547 Injection in the Treatment of Subjects With Super-Refractory Status Epilepticus
Brief Title: A Study With SAGE-547 for Super-Refractory Status Epilepticus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 547-SSE-301
Record Dates: First submitted 2015-06-02; First posted 2015-06-23 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2022-01

CONDITIONS: Super-Refractory Status Epilepticus
MeSH Terms: interventions — brexanolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAGE-547 (Active Comparator): Intravenous
  Interventions: Drug: SAGE-547
- Placebo (Placebo Comparator): Intravenous
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAGE-547
  Arms: SAGE-547
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial, designed to evaluate the efficacy and safety of SAGE-547 administered as a continuous intravenous infusion to subjects in Super-Refractory Status Epilepticus (SRSE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects two (2) years of age and older
* Subjects who have:

  * Failed to respond to the administration of at least one first-line agent (e.g., benzodiazepine or other emergent initial anti-epileptic drug [AED] treatment), according to institution standard of care, and;
  * Failed to respond to at least one second-line agent (e.g., phenytoin, fosphenytoin, valproate, phenobarbital, levetiracetam or other urgent control AED), according to institution standard of care, and;
  * Not previously been administered a third-line agent but have been admitted to an intensive care unit with the intent of administering at least one third-line agent for at least 24 hours; or who have previously failed zero, one or more wean attempts from third-line agents and are now on continuous intravenous infusions of one or more third-line agent and in an EEG burst or seizure suppression pattern; or who have previously failed one or more wean attempts from third-line agents and are now either not on a continuous intravenous infusion of at least one third-line agent or are on a continuous intravenous infusion of one or more third-line agent but not in an EEG burst or seizure suppression pattern

Exclusion Criteria:

* Subjects with SRSE due to anoxic/hypoxic encephalopathy with highly malignant/ malignant EEG features
* Children (subjects aged less than 17 years) with an encephalopathy due to a rapidly progressing underlying neurological disorder
* Subjects who have any of the following:

  1. a glomerular filtration rate (GFR) low enough to warrant dialysis but for whatever reason, dialysis is not planned or non-continuous dialysis planned (that would not adequately remove Captisol®);
  2. severe cardiogenic or vasodilatory shock requiring two or more pressors that is not related to third-line agent use;
  3. fulminant hepatic failure;
  4. no reasonable expectation of recovery (for instance, a likely outcome is persistent vegetative state) or life-expectancy, in the experience of the investigator, is less than 30 days.
* Subjects who are being administered more than three third-line agents concomitantly or in whom the qualifying wean cannot be completed per protocol

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07-18 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rosenthal, MD, Principal Investigator — Massachusetts General Hospital; Mark Wainwright, MD, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (137):
- United States (79):
  - Sage Investigational Site, Birmingham, Alabama
  - Sage Investigational Site, Mobile, Alabama
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, Fresno, California
  - Sage Investigational Site, Loma Linda, California
  - Sage Investigational Site, Los Angeles, California
  - Sage Investigational Site, Roseville, California
  - Sage Investigational Site, Sacramento, California
  - Sage Investigational Site, New Haven, Connecticut
  - Sage Investigational Site, Wilmington, Delaware
  - Sage Investigational Site, Washington D.C., District of Columbia
  - Sage Investigational Site, Gainesville, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Sarasota, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Weston, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Honolulu, Hawaii
  - Sage Investigational Site, Boise, Idaho
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Maywood, Illinois
  - Sage Investigational Site, Peoria, Illinois
  - Sage Investigational Site, Springfield, Illinois
  - Sage Investigational Site, Urbana, Illinois
  - Sage Investigational Site, Iowa City, Iowa
  - Sage Investigational Site, Wichita, Kansas
  - Sage Investigational Site, Lexington, Kentucky
  - Sage Investigational Site, Louisville, Kentucky
  - Sage Investigational Site, Baton Rouge, Louisiana
  - Sage Investigational Site, New Orleans, Louisiana
  - Sage Investigational Site, Portland, Maine
  - Sage Investigational Site, Baltimore, Maryland
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Newton, Massachusetts
  - Sage Investigational Site, Ann Arbor, Michigan
  - Sage Investigational Site, Detroit, Michigan
  - Sage Investigational Site, East Lansing, Michigan
  - Sage Investigational Site, Grand Rapids, Michigan
  - Sage Investigational Site, Royal Oak, Michigan
  - Sage Investigational Site, Minneapolis, Minnesota
  - Sage Investigational Site, Rochester, Minnesota
  - Sage Investigational Site, Jackson, Mississippi
  - Sage Investigational Site, Kansas City, Missouri
  - Sage Investigational Site, St Louis, Missouri
  - Sage Investigational Site, Edison, New Jersey
  - Sage Investigational Site, Morristown, New Jersey
  - Sage Investigational Site, New Brunswick, New Jersey
  - Sage Investigational Site, Summit, New Jersey
  - Sage Investigational Site, Buffalo, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Port Jefferson, New York
  - Sage Investigational Site, Rochester, New York
  - Sage Investigational Site, Syracuse, New York
  - Sage Investigational Site, Durham, North Carolina
  - Sage Investigational Site, Winston-Salem, North Carolina
  - Sage Investigational Site, Akron, Ohio
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Cleveland, Ohio
  - Sage Investigational Site, Columbus, Ohio
  - Sage Investigational Site, Toledo, Ohio
  - Sage Investigational Site, Portland, Oregon
  - Sage Investigational Site, Hershey, Pennsylvania
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Pittsburgh, Pennsylvania
  - Sage Investigational Site, Charleston, South Carolina
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Nashville, Tennessee
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Dallas, Texas
  - Sage investigational Site, San Antonio, Texas
  - Sage Investigational Site, Salt Lake City, Utah
  - Sage Investigational Site, Burlington, Vermont
  - Sage Investigational Site, Seattle, Washington
  - Sage Investigational Site, Huntington, West Virginia
  - Sage Investigational Site, Morgantown, West Virginia
  - Sage Investigational Site, Wauwatosa, Wisconsin
- Austria (2):
  - Sage Investigational Site, Innsbruck
  - Sage Investigational Site, Salzburg
- Canada (5):
  - Sage Investigational Site, Vancouver, British Columbia
  - Sage Investigational Site, Hamilton, Ontario
  - Sage Investigational Site, Kingston, Ontario
  - Sage Investigational Site, London, Ontario
  - Sage Investigational Site, Montreal, Quebec
- Sage Investigational Site, Copenhagen, Denmark
- Estonia (2):
  - Sage Investigational Site, Tallinn
  - Sage Investigational Site, Tartu
- Finland (2):
  - Sage Investigational Site, Helsinki
  - Sage Investigational Site, Kuopio
- France (6):
  - Sage Investigational Site, Bron
  - Sage Investigational Site, Dijon
  - Sage Investigational Site, Lille
  - Sage Investigational Site, Limoges
  - Sage Investigational Site, Lyon
  - Sage Investigational Site, Paris
- Germany (3):
  - Sage Investigational Site, Hamburg
  - Sage Investigational Site, Marburg
  - Sage Investigational Site, Osnabrück
- Hungary (2):
  - Sage Investigational Site, Balassagyarmat
  - Sage Investigational Site, Budapest
- Israel (6):
  - Sage Investigational Site, Ashkelon
  - Sage Investigational Site, Holon
  - Sage Investigational Site, Jerusalem
  - Sage Investigational Site, Petah Tikva
  - Sage Investigational Site, Tel Litwinsky
  - Sage Investigational Site, Tzrifin
- Italy (9):
  - Sage Investigational Site, Bologna
  - Sage Investigational Site, Florence
  - Sage Investigational Site, Milan
  - Sage Investigational Site, Modena
  - Sage Investigational Site, Monza
  - Sage Investigational Site, Perugia
  - Sage Investigational Site, Reggio Calabria
  - Sage Investigational Site, Rome
  - Sage Investigational Site, Verona
- Netherlands (4):
  - Sage Investigational Site, Enschede
  - Sage Investigational Site, Heerlen
  - Sage Investigational Site, Maastricht
  - Sage Investigational Site, Nijmegen
- Serbia (3):
  - Sage Investigational Site, Belgrade
  - Sage Investigational Site, Niš
  - Sage Investigational Site, Novi Sad
- Spain (7):
  - Sage Investigational Site, Badalona
  - Sage Investigational Site, Barakaldo
  - Sage Investigational Site, Barcelona
  - Sage Investigational Site, Córdoba
  - Sage Investigational Site, Granada
  - Sage Investigational Site, L'Hospitalet de Llobregat
  - Sage Investigational Site, Madrid
- Sage Investigational Site, Gothenburg, Sweden
- United Kingdom (5):
  - Sage Investigational Site, Manchester
  - Sage Investigational Site, Norfolk
  - Sage Investigational Site, Norwich
  - Sage Investigational Site, Staffordshire
  - Sage Investigational Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- See also: Sage Therapeutics — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 122 investigative sites in Canada, United States, Austria, Denmark, Estonia, Finland, France, Germany, Israel, Italy, Serbia, Spain and United Kingdom from 31 July 2015 to 11 August 2017.
Pre-assignment Details: Participants 2 years of age and older with Super-Refractory Status Epilepticus were eligible. One participant in the placebo group was erroneously given SAGE-547 and was, therefore, included in the SAGE- 547 group.
Groups:
- Placebo: Placebo was administered over the course of 6 days, beginning with a 1-hour dose rate equivalent to 300 micrograms per kilogram per hour (μg/kg/h) of the active arm loading dose, followed by a maintenance period achieving a maximum of 90 μg/kg/h (double-blind treatment), which included a step-wise taper during the last 24 hours of treatment.
- SAGE-547: SAGE-547 Injection was administered over the course of 6 days, beginning with a 1-hour 300 μg/kg/h loading dose, followed by a maintenance period achieving a maximum of 90 μg/kg/h (double-blind treatment) or 150 μg/kg/h (open-label treatment), both of which included a step-wise taper during the last 24 hours of treatment. Eligible participants, who did not respond to blinded study treatment, were allowed to enter an Open-label Treatment Period of identical duration.
Period: Overall Study
Arm/Group | Placebo | SAGE-547
Started | 65 | 67
Intent-to-Treat Analysis Set | 66 | 66
Completed (Participants who completed both study drug and study visits.) | 50 | 53
Not Completed | 15 | 14
Not completed — Completed Visits but Discontinued Drug | 2 | 1
Not completed — Died in Double-Blind Treatment Period | 11 | 11
Not completed — Adverse Event | 1 | 1
Not completed — Transferred Away from Study Site | 1 | 0
Not completed — Left Study Site for Rehabilitation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who had an infusion of blinded study drug initiated. One participant in the placebo group was erroneously given SAGE-547 and was, therefore, included in the SAGE-547 group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-547 | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (22.69) | 41.3 (23.89) | 39.6 (23.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 35 | 32 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 45 | 92
  Black | 14 | 13 | 27
  Asian | 3 | 5 | 8
  Other | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 55 | 61 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Able to be Weaned Off All Third-Line Agents Prior to End of Double-Blind SAGE-547 or Placebo Infusion, and Remain Off All Third-Line Agents for ≥ 24 Hours Following the End of SAGE-547 or Placebo Infusion
Description: Third-line agents were anesthetic agents that were administered in order to reach a seizure or burst suppression electroencephalogram (EEG) pattern. For this study, third-line agents were defined as continuous intravenous infusions of pentobarbital/thiopental, midazolam, propofol, and ketamine at maintenance doses alone or in combination sufficient to produce a burst or seizure suppression pattern on the EEG. A responder was a participant who was able to be weaned off all third-line agents prior to the end of the SAGE-547 or placebo infusion and remain off all third-line agents for >=24 hours after the end of the study drug infusion. The primary analysis was a comparison between SAGE-547 and placebo of the proportion of responders.
Time Frame: 7 days
Population: The Intent-to-Treat Analysis Set included all participants who had an infusion of blinded study drug initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
Participants | 28 | 29
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.878, Regression, Logistic; Odds Ratio (OR) = 1.056, 95% CI 2-sided [0.527 to 2.118]

2. Secondary Outcome: Time Between the Primary Outcome Response and the Re-institution of Any Third-line Agent for Seizure or Burst Suppression
Description: Third-line agents were anesthetic agents that were administered in order to reach a seizure or burst suppression EEG pattern. For this study, third-line agents were defined as continuous intravenous infusions of pentobarbital/thiopental, midazolam, propofol, and ketamine at maintenance doses alone or in combination sufficient to produce a burst or seizure suppression pattern on the EEG. A responder was a participant who was able to be weaned off all third-line agents prior to the end of the SAGE-547 or placebo infusion and remain off all third-line agents for >=24 hours after the end of the study drug infusion. The primary analysis was a comparison between SAGE-547 and placebo of the proportion of responders.
Time Frame: Up to 21 days
Population: The Intent-to-Treat Analysis Set included all participants who had an infusion of blinded study drug initiated. Here, overall number of participants analyzed (N) indicates participants analyzed for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 28 | 29
days | 13.500 [0.06 to 18.00] | 14.000 [0.18 to 16.00]
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.636, Regression, Cox; Hazard Ratio (HR) = 0.747, 95% CI 2-sided [0.222 to 2.507]

3. Secondary Outcome: Number of Participants Able to be Weaned Off All Third-line Agents Before the End of the First SAGE-547 or Placebo Infusion
Description: Third-line agents were anesthetic agents that were administered in order to reach a seizure or burst suppression EEG pattern. For this study, third-line agents were defined as continuous intravenous infusions of pentobarbital/thiopental, midazolam, propofol, and ketamine at maintenance doses alone or in combination sufficient to produce a burst or seizure suppression pattern on the EEG.
Time Frame: Day 6
Population: The Intent-to-Treat Analysis Set included all participants who had an infusion of blinded study drug initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
Participants | 45 | 38
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.199, Regression, Logistic; Odds Ratio (OR) = 0.623, 95% CI 2-sided [0.303 to 1.282]

4. Secondary Outcome: Time Between the Secondary Outcome Measure Response and the Re-institution of Any Third-line Agent for Seizure or Burst Suppression
Description: as for outcome 3
Time Frame: Up to 21 days
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 45 | 38
days | 7.000 [0.00 to 20.00] | 15.000 [0.00 to 19.00]
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.328, Regression, Cox; Hazard Ratio (HR) = 0.683, 95% CI 2-sided [0.318 to 1.466]

5. Secondary Outcome: Change in Clinical Global Impression Scale (CGI)
Description: The CGI scale was used to integrate several sources of information into a single rating of a participant's condition. The CGI was rated on a 7-point scale, from a minimum of 0 to a maximum of 7, where 0 = Not assessed; 1 = Normal, not at all ill; 2 = Borderline physically ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill participants. A negative change from baseline indicates improvement. A positive change from baseline indicates worsening. Here, study visits followed by "R" indicate the Open-label Treatment Period.
Time Frame: Up to 21 days
Population: The Intent-to-Treat Analysis Set included all participants who had an infusion of blinded study drug initiated. Here, number of participants analyzed (N) indicates participants with available data at each time point for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
units on scale
  Baseline: number analyzed (Participants) | 66 | 65
  Baseline | 6.0 (0.89) | 5.9 (1.31)
  Visit 12: number analyzed (Participants) | 33 | 32
  Visit 12 | -1.0 (1.42) | -0.6 (1.91)
  Visit 12R: number analyzed (Participants) | 18 | 20
  Visit 12R | -0.7 (1.36) | -0.5 (1.19)

6. Secondary Outcome: Number of Days After the End of the First Study Drug Infusion Without Status Epilepticus, Up to Visit 12
Description: Here, study visits followed by "R" indicate the Open-label Treatment Period.
Time Frame: Up to 21 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
days
  Visit 12: number analyzed (Participants) | 41 | 40
  Visit 12 | 10.05 (6.738) | 11.15 (6.058)
  Visit 12R: number analyzed (Participants) | 25 | 26
  Visit 12R | 11.08 (6.557) | 9.23 (6.345)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.339, Regression, Cox; Hazard Ratio (HR) = 0.583, 95% CI 2-sided [0.193 to 1.763]

7. Secondary Outcome: Number of Days After the End of the First Study Drug Infusion Without Seizures (Convulsive and Non-convulsive), up to Visit 12
Description: Here, study visits followed by "R" indicate the Open-label Treatment Period.
Time Frame: Up to 21 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
days
  Visit 12: number analyzed (Participants) | 41 | 40
  Visit 12 | 8.22 (7.289) | 7.50 (6.626)
  Visit 12R: number analyzed (Participants) | 25 | 26
  Visit 12R | 7.52 (7.054) | 6.08 (5.932)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.817, Regression, Cox; Hazard Ratio (HR) = 1.086, 95% CI 2-sided [0.539 to 2.189]

8. Secondary Outcome: Number of Separate Episodes of Status Epilepticus Up to Visit 12
Description: Here, study visits followed by "R" indicate the Open-label Treatment Period.
Time Frame: Up to 21 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
episodes
  Visit 12: number analyzed (Participants) | 9 | 5
  Visit 12 | 1.3 (0.50) | 1.4 (0.55)
  Visit 12R: number analyzed (Participants) | 5 | 8
  Visit 12R | 2.2 (2.17) | 1.0 (0.00)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547; Test type: Superiority; p = 0.567, ANCOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.9 to 0.5]

9. Secondary Outcome: Number of Participants With a New Diagnosis of Epilepsy After Visit 11
Description: Here, study visits followed by "R" indicate the Open-label Treatment Period.
Time Frame: Up to 21 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-547
Number analyzed (Participants) | 66 | 66
Participants
  Visit 12: number analyzed (Participants) | 34 | 34
  Visit 12 | 0 | 5
  Visit 12R: number analyzed (Participants) | 20 | 23
  Visit 12R | 5 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 27 days
Description: The Safety Analysis Set included all subjects who had an infusion of blinded study drug initiated.
Arm/Group | Placebo | SAGE-547
All-Cause Mortality (participants affected / at risk) | 12/65 | 17/67
Serious Adverse Events (participants affected / at risk) | 22/65 | 27/67
Other Adverse Events (participants affected / at risk) | 58/65 | 60/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | SAGE-547 (N=67)
Cardiac arrest (Cardiac disorders) | 4 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block (Cardiac disorders) | 0 | 1
Torsade de pointes (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Mitochondrial DNA mutation (Congenital, familial and genetic disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 2 | 0
Mydriasis (Eye disorders) | 1 | 0
Pupil fixed (Eye disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Device related thrombosis (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Septic shock (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Serratia sepsis (Infections and infestations) | 1 | 0
Subdural empyema (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Brain herniation (Injury, poisoning and procedural complications) | 3 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Propofol infusion syndrome (Metabolism and nutrition disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 2
Status epilepticus (Nervous system disorders) | 2 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Withdrawal of life support (Surgical and medical procedures) | 7 | 11
Hypotension (Vascular disorders) | 1 | 2
Neurogenic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | SAGE-547 (N=67)
Anaemia (Blood and lymphatic system disorders) | 7 | 12
Leukocytosis (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 3
Tachycardia (Cardiac disorders) | 4 | 8
Atrial fibrillation (Cardiac disorders) | 2 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 12
Constipation (Gastrointestinal disorders) | 8 | 10
Vomiting (Gastrointestinal disorders) | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Pyrexia (General disorders) | 21 | 19
Hyperthermia (General disorders) | 1 | 5
Peripheral swelling (General disorders) | 0 | 4
Oedema (General disorders) | 4 | 3
Hypothermia (General disorders) | 4 | 1
Urinary tract infection (Infections and infestations) | 14 | 13
Pneumonia (Infections and infestations) | 11 | 13
Fungal infection (Infections and infestations) | 1 | 4
Sepsis (Infections and infestations) | 4 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 5
Lipase increased (Investigations) | 6 | 5
Alanine aminotransferase increased (Investigations) | 5 | 4
Blood potassium decreased (Investigations) | 1 | 4
White blood cell count increased (Investigations) | 0 | 4
Electrocardiogram QT prolonged (Investigations) | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 8
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 8
Hypernatraemia (Metabolism and nutrition disorders) | 6 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 5
Fluid overload (Metabolism and nutrition disorders) | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 3
Agitation (Psychiatric disorders) | 4 | 5
Haematuria (Renal and urinary disorders) | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 8 | 5
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Hypertension (Vascular disorders) | 6 | 8
Hypotension (Vascular disorders) | 10 | 6
Deep vein thrombosis (Vascular disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT02477618/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT02477618/SAP_000.pdf